CLINICAL TRIAL: NCT03808545
Title: Comprehensive Lifestyle Intervention for Reducing Cardiometabolic Risk and Symptom Burden in Adults With Multiple Sclerosis
Brief Title: Activity and Balanced Eating to Reduce Comorbidities and Symptoms of MS
Acronym: ABC's of MS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brooks C. Wingo, PhD, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300002096; P30DK056336 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2019-01-17 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Behavior Therapy; Exercise; Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIPAMS (Active Comparator): All participants will receive the standard BIPAMS intervention for the first 8 weeks of the trial.Those in the BIPAMS group will continue receiving the established BIPAMS intervention for the remainder of the trial.
  Interventions: Behavioral: Behavioral Intervention for Physical Activity in Multiple Sclerosis (BIPAMS)
- BIPAMS + Diet (Experimental): All participants will receive the standard BIPAMS intervention for the first 8 weeks of the trial.Those in the BIPAMS+Diet arm will begin receiving dietary materials in week 9.
  Interventions: Behavioral: BIPAMS + Diet

INTERVENTIONS:
Behavioral: Behavioral Intervention for Physical Activity in Multiple Sclerosis (BIPAMS) — This is a newly developed Internet website that delivered a Social Cognitive Theory-based behavioral intervention using e-learning and one-on-one video chats approaches for increasing physical activity and improving symptoms, walking impairment, and neurological disability. The intervention will last 16 weeks and will include physical activity information.
  Arms: BIPAMS
Behavioral: BIPAMS + Diet — For 8 weeks a participant will complete the standard BIPAMS intervention. For the subsequent 8 weeks, in addition to the BIPAMS website, participants will receive a diet prescription with instructions and guidance on their one-on-one video calls and will utilize the HealthWatch360 app and/or desktop website to track their dietary intake. The total intervention will last 16 weeks and will include physical activity information and dietary information.
  Arms: BIPAMS + Diet

SUMMARY:
Multiple sclerosis (MS) is the leading cause of irreversible neurological disability among young women and the second leading cause of disability among young men in the U.S. Cardiometabolic risk factors including obesity and hyperlipidemia are common among people with MS, and these risk factors are associated with severity and frequency of MS relapses and disease progression. People with MS often experience symptoms of pain, fatigue, and depression, which make adhering to a healthy lifestyle difficult, as evidenced by the high rates of unhealthy behaviors including poor diet and physical inactivity among this group. Physical activity has reduced symptoms of MS and improved metabolic risk profiles, but little research has focused on the role of a dietary intervention combined with physical activity in this group. Therefore, the purpose of this study is to test the efficacy of a combined diet and physical activity intervention for reducing cardiometabolic risks and MS symptoms when compared to a physical activity intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-Remitting MS
* On disease modifying treatment for 6 months
* No relapse within the previous 30 days
* BMI 25-55 kg/m2
* Self-identify as not currently meeting recommendations for healthy diet and physical activity
* Ambulatory with or without assistance
* Reliable access to the internet via computer or smartphone
* Responsible for their personal food preparation or have input into the food prepared for them
* Score indicating low cognitive functioning on the Telephone Interview for Cognitive Status assessment

Exclusion Criteria:

* Physician does not approve participation
* Use of the following diabetes medications: Acetohexamide, Chlorpropamide (Diabinese), Tolbutamide (Orinase, Tol-Tab), Tolazamide (Tolinase), Glipizide (Glucotrol, Glucotrol XL, Metaglip), Glyburide (Micronase, DiaBeta, Glynase, Glucovance), Glimepiride (Amaryl), Humalog or lispro, Novolog or aspart, Apidra or glulisine, Regular (R) humulin or novolin, Velosulin (for use in the insulin pump), NPH (N), Lente (L), Ultralente (U), Lantus, Levemir or detemir, Humulin 70/30, Novolin 70/30, Novolog 70/30, Humulin 50/50, or Humalog mix 75/25
* Already on a specific diet meant to improve health
* Heart attack, stroke, or heart bypass surgery less than 6 months ago
* Pulmonary disease, cardiovascular disease or renal failure less than 6 months ago
* Smoking
* Cancer, HIV or liver/kidney disease
* Inability to travel to Lakeshore for testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeshore Foundation, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIPAMS | BIPAMS + Diet
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Only study completers were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | BIPAMS | BIPAMS + Diet | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants] — Population: Only completers were analyzed.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 4 | 9
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only study completers were analyzed.
  Participants
    Female | 5 | 3 | 8
    Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only study completers were analyzed.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 3 | 5
    White | 3 | 1 | 4
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: BMI Change
Description: BMI will be calculated using the formula weight/height2 (kg/m^2). Height will be measured with participants standing against the wall. Weight will be assessed using a digital scale. BMI change will be calculated the difference between 16 week BMI and baseline BMI.
Time Frame: Baseline and16 weeks
Population: Only study completers were analyzed.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
kg/m2 | .60 (1.36) | .49 (1.30)

2. Primary Outcome: Waist Circumference Change
Description: Waist circumference will be measured twice at the level of the umbilicus after normal expiration, with the participant standing. If the two values differ by >1 cm, a third measurement will be taken and the results of the two or three trials averaged. Waist circumference change will be calculated as the difference between 16 week waist circumference and baseline waist circumference.
Time Frame: Baseline and 16 weeks
Population: Study completers
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
cm | .31 (3.07) | .31 (5.54)

3. Primary Outcome: Fat Mass Change
Description: Participants will undergo a total body scan measuring total body composition on a Lunar iDXA with enCORE software version 13.6 (GE Healthcare, Chicago, IL). Fat mass (FM) change will be calculated the difference between 16 week FM and baseline FM.
Time Frame: Baseline and 16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
lb | 2.14 (6.07) | .05 (3.07)

4. Secondary Outcome: Diastolic Blood Pressure Change
Description: Diastolic blood pressure (DBP) will be obtained using a sphygmomanometer. DBP will be measured twice, with a resting time of 1 minute in between each measurement. The results of the two trials will be averaged. DBP change will be calculated as the difference between 16 week DBP and baseline DBP.
Time Frame: Baseline and 16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
mmHG | -2.20 (9.60) | .00 (5.72)

5. Secondary Outcome: Systolic Blood Pressure Change
Description: Systolic blood pressure (BP) will be obtained using a sphygmomanometer. SBP will be measured twice, with a resting time of 1 minute in between each measurement. The results of the two trials will be averaged. SBP change will be calculated as the difference between 16 week SBP and baseline SBP.
Time Frame: Baseline and 16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
mmHg | -6.20 (8.93) | -4.25 (14.77)

6. Secondary Outcome: Glucose Change
Description: Two (2) vials of blood will be drawn (7 mL or 1.4 teaspoons) via venipuncture. Glucose, along with other blood measures, will be assessed from this blood sample. Glucose change will be calculated as the difference between 16 week glucose and baseline glucose.
Time Frame: Baseline and16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
mg/dl | -3.40 (7.67) | .00 (14.31)

7. Secondary Outcome: Insulin Change
Description: Two (2) vials of blood will be drawn (7 mL or 1.4 teaspoons) via venipuncture. Insulin, along with other blood measures, will be assessed from this blood sample. Insulin change will be calculated the difference between 16 week insulin and baseline insulin.
Time Frame: Baseline and16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: microUnits/mL
Groups:
- BIPAMS: All participants will receive the standard BIPAMS intervention for the first 8 weeks of the trial. Those in the BIPAMS group will continue receiving the established BIPAMS intervention for the remainder of the trial.
  Behavioral Intervention for Physical Activity in Multiple Sclerosis (BIPAMS): This is a newly developed Internet website that delivered a Social Cognitive Theory-based behavioral intervention using e-learning and one-on-one video chats approaches for increasing physical activity and improving symptoms, walking impairment, and neurological disability. The intervention will last 16 weeks and will include physical activity information.
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
microUnits/mL | -2.76 (4.00) | -2.80 (11.14)

8. Secondary Outcome: Triglycerides Change
Description: Two (2) vials of blood will be drawn (7 mL or 1.4 teaspoons) via venipuncture. Triglycerides, along with other blood measures, will be assessed from this blood sample. Triglyceride change will be calculated as the difference between 16 week triglycerides and baseline triglycerides.
Time Frame: Baseline and 16 weeks
Population: Completers only; BIPAMS group outlier lab value (n=1) was excluded from analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 4 | 4
mg/dl | 4.50 (14.20) | -12.50 (14.53)

9. Secondary Outcome: LDL-C Change
Description: Two (2) vials of blood will be drawn (7 mL or 1.4 teaspoons) via venipuncture. LDL-C, along with other blood measures, will be assessed from this blood sample. LDL-C change will be calculated as the difference between 16 week LDL-C and baseline LDL-C.
Time Frame: Baseline and16 weeks
Population: Completers only; BIPAMS group outlier lab value (n=1) was excluded from analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 4 | 4
mg/dl | -17.40 (5.97) | 10.50 (20.69)

10. Secondary Outcome: HDL-C Change
Description: Two (2) vials of blood will be drawn (7 mL or 1.4 teaspoons) via venipuncture. HDL-C, along with other blood measures, will be assessed from this blood sample. HDL-C change will be calculated the difference between 16 week HDL-C and baseline HDL-C.
Time Frame: Baseline and 16 weeks
Population: Only completers were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
mg/dL | -6.40 (6.95) | 1.00 (7.44)

11. Secondary Outcome: Total Cholesterol Change
Description: Two (2) vials of blood will be drawn (7 mL or 1.4 teaspoons) via venipuncture. Total cholesterol (TC), along with other blood measures, will be assessed from this blood sample. TC change will be calculated as the difference between 16 week TC and baseline TC.
Time Frame: Baseline and 16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
mg/dl | -12.00 (19.81) | 9.00 (29.47)

12. Secondary Outcome: Change in Fatigue Severity Scale
Description: Measured by the Fatigue Severity Scale (FSS). The total score is the sum of the 9 items. The range for scoring is 9-63, with higher scores indicating greater fatigue severity. Change in fatigue will be calculated as the difference between 16-week FSS and baseline FSS.
Time Frame: Baseline and16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
score on a scale | 1.20 (5.63) | 4.00 (9.24)

13. Secondary Outcome: Change in Modified Fatigue Impact Scale
Description: Measured by the Modified Fatigue Impact Scale (MFIS). The total score is the sum of the 5 items. The range for scoring is 0-20, with higher scores indicating greater fatigue. Change in fatigue will be calculated as the difference between 16-week MFIS and baseline MFIS.
Time Frame: Baseline and 16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
score on a scale | .40 (7.57) | -2.50 (13.72)

14. Secondary Outcome: Change in Depression Symptoms
Description: Measured by the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, divided into two 7 item subscales. The total score is the sum of the 7 items from each subscale, and ranges from 0- 21 for the depression subscale. Higher scores in the depression subscale questions indicates greater levels of depression. Change in depression symptoms will be calculated as the difference between 16-week HADS depression subscale and baseline HADS depression subscale.
  Minimum score: 0; Maximum Score Depression subscale: 21
Time Frame: Baseline and 16 weeks
Population: Completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
score on a scale | 2.40 (2.19) | .25 (.96)

15. Secondary Outcome: Change in Anxiety
Description: Measured by the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, divided into two 7 item subscales. The total score is the sum of the 7 items from each subscale, and ranges from 0- 21 for the anxiety subscale. Higher scores in the anxiety subscale questions indicates greater levels of anxiety. Change in anxiety will be calculated as the difference between 16-week HADS anxiety subscale and baseline HADS anxiety subscale.
  Minimum score: 0; Maximum score anxiety subscale: 21
Time Frame: Baseline and16 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIPAMS | BIPAMS + Diet
Number analyzed (Participants) | 5 | 4
score on a scale | 0.40 (2.61) | -2.00 (1.41)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: All hospitalizations are included, regardless of reason or relation to study participation.
Arm/Group | BIPAMS | BIPAMS + Diet
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIPAMS (N=6) | BIPAMS + Diet (N=5)
Hospitalization (Nervous system disorders) | 0 (0) | 1 (1) — Participant was hospitalized for MS relapse.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIPAMS (N=6) | BIPAMS + Diet (N=5)
Elevated blood pressure (Cardiac disorders) | 0 (0) | 1 (1) — Participant reported elevated blood pressure for 2 weeks.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Early termination was due to inability to recruit sufficient participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03808545/Prot_SAP_ICF_000.pdf